CLINICAL TRIAL: NCT05326321
Title: Effect of Virtual Reality Headset Glasses Used in The Arteriovenous Fistule Cannulation Processon Paın and Patient Satisfaction
Brief Title: Effect of Virtual Reality Glasses in The Arteriovenous Fistule Cannulation Processon Paın and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Didem Lafci, PhD, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Mersin Universi
Record Dates: First submitted 2022-03-25; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Arteriovenous Fistula
Keywords: Virtual Reality Glasses; Nursing; Pain; Patient Satisfaction
MeSH Terms: conditions — Arteriovenous Fistula; Pain; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm, randomized controlled clinical trial
Who Masked: Participant
Masking Description: According to the randomization table, the information showing the patients included in the research sample is assigned to the A and B groups will be put in an opaque envelope. This envelope will be kept by the coordinator researcher (DL) and when the researcher (HŞ) goes to the patient for application, after filling out the "Informed Voluntary Consent Form", he will open the envelope and learn which group is in which group. Due to the nature of the study, patients and the researcher (HŞ) will not be blinded, since abdominal massage will be applied only to the patients included in the study. When the research is completed, the data will be transferred to the computer environment by a statistician who does not know the A and B groups, and the data will be analyzed by a statistician independent of the research and the findings will be reported. Thus, the data analysis and statistics phase will be blind to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Glasses Group (Experimental): The patients in the intervention group were shown a video with virtual reality glasses for an average of 5 minutes, 2 minutes before the start of the AVF cannulation procedure and 3 minutes throughout the procedure. After the AVF cannulation procedure was completed and 10 minutes later, the VAS and Hemodynamic Variables Follow-up Form were reapplied, and the 2nd and 3rd measurements were obtained. Patients' satisfaction was measured with VAS 10 minutes after the procedure. During the application of virtual reality glasses, a screen was pulled between the patients in the intervention and control groups so that there would be no interaction.
  Interventions: Other: Study Group
- Control group (No Intervention): Without any application to the patients in the control group, the AVF cannulation procedure before HD was performed with the constant site-area puncture technique used by the clinic (after the patient was placed in the fowler position, the arterial needle was 3 cm away from the anastomosis at an angle of 20°-45° towards the distal, and the venous needle was from the arterial needle. 3-5 cm more proximal, again at an angle of 20°-45°) was performed by the HD nurse. The 1st, 2nd and 3rd measurements were obtained as in the intervention group.

INTERVENTIONS:
Other: Study Group — The patients in the intervention group were shown a video with virtual reality glasses for an average of 5 minutes, 2 minutes before the start of the AVF cannulation procedure and 3 minutes throughout the procedure.
  Arms: Virtual Reality Glasses Group

SUMMARY:
This research was conducted as a randomized controlled experimental study aiming to determine the impact of virtual reality glasses used in the AVF process on the pain felt by patients and patient satisfaction.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a progressive, irreversible renal disease in which the ability of the body to maintain the balance of metabolism, fluid and electrolytes fails. Chronic kidney disease (CKD) is one of the major health problems with an increasing prevalence in the World. Hemodialysis as one of the most common methods of renal replacement therapy is a stressful procedure despite to maintain the survival of patients with chronic kidney disease that permanent and safe vascular access is one of the requirements of a successful hemodialysis. The pain of AVF puncture is common among the patients undergoing HD as acute and chronic pain which reported in more than 82% and 92% of them, respectively. Experience of the arteriovenous fistula puncture-related pain can have unpleasant effects on the patients, it causes that hemodialysis patients experience more disability, depression, irritability, and insomnia than other patients in adapting to stress. Experiencing continued pain can also affect the level of hemodialysis acceptance in patients and ultimately decrease quality of life. Therefore, pain control is an important priority in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Receiving HD treatment
* Open to communication
* Fully oriented
* Without vision, hearing and perception problems
* Without any psychiatric illness
* Without a history of seizures such as epilepsy
* HD treatment administered via AVF
* İn the last day, no injection was made into any artery or vein from the place where the intervention will be performed
* Without any signs of infection such as redness, swelling, open wound in the area where the intervention will be performed
* Standardized Mini Mental Test value is 24 points and above
* One-time needle attempt from AV

Exclusion Criteria:

* Refusing to participate in the study
* under the age of 18
* Can't speak Turkish
* Closed to communication and not fully oriented
* Visual, hearing and perception problems
* Any psychiatric illness
* Having a history of seizures such as epilepsy
* HD treatment not administered via AVF
* Injection into any artery or vein from the place where the intervention will be performed in the last day,
* Any signs of infection such as redness, swelling, open wound in the area to be operated
* Using any pain medication before the procedure on the same day
* SMMT value below 24 in patients over 65 years of age
* Cannulation procedure not performed with a 16 G AVF needle
* Patients with multiple injections from the AVF

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

PRIMARY OUTCOMES:
Pain evaluated using the Visual Analog Scale | Change from before implementation, immediately after the procedure and after 10 minutes of practice (Virtual Reality Headset Glasses)
  The patient marks a value between 1 and 10 on the Visual Analog Scale (VAS). As the value increases, the severity of pain increases.

SECONDARY OUTCOMES:
Blood pressure | Change from before implementation, immediately after the procedure and after 10 minutes of practice (Virtual Reality Headset Glasses)
  systolic blood pressure (SBP), diastolic blood pressure (DBP), mmHg
Heart rate | Change from before implementation, immediately after the procedure and after 10 minutes of practice (Virtual Reality Headset Glasses)
  beats per minute
respiratory rate | Change from before implementation, immediately after the procedure and after 10 minutes of practice (Virtual Reality Headset Glasses)
  ekspiration and inspiration per minute
peripheral oxygen saturation | Change from before implementation, immediately after the procedure and after 10 minutes of practice (Virtual Reality Headset Glasses)
  %, percentage of oxygenated hemoglobin in peripheral arterial blood

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Şen, Master, Principal Investigator — Pozantı State Hospital
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No